CLINICAL TRIAL: NCT00593515
Title: Effects of Parental Behavior on Child Anxiety Regulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Jeffrey J. Wood, UCLA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1F31MH064999 (NIH)
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Separation Anxiety Disorder; Social Phobia; Generalized Anxiety Disorder
MeSH Terms: conditions — Anxiety, Separation; Phobia, Social; Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Family CBT
  Interventions: Behavioral: Family cognitive behavioral therapy
- 2 (Active Comparator): Child-focused CBT
  Interventions: Behavioral: Child-focused cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Family cognitive behavioral therapy — 12-16 weekly sessions of family cognitive behavioral therapy, 60-80 minutes each
  Arms: 1
Behavioral: Child-focused cognitive behavioral therapy — 12-16 weekly sessions of child-focused cognitive behavioral therapy, 60-80 minutes each
  Arms: 2

SUMMARY:
Does parenting style affect emotion regulation among children who initially demonstrate high levels of fear and anxiety? Although recent correlational research has demonstrated a linkage between parental behaviors, such as excessive intrusiveness, and children's manifestations of fear and anxiety, it is not clear if parenting behaviors directly influence children's ability to regulate these emotions. Alternatively, these parental behaviors may be elicited by children who express fears and anxieties more frequently than other children do. Experimental research designs would offer a more definitive test of these competing explanations of the extant correlational findings. Intervention studies, in particular, can test whether experimentally manipulating current family interaction patterns affects children's ability to regulate emotion. This study provides a preliminary experimental test of the relationship between parental behavior and children's regulation of fear and anxiety. Some 40 clinically anxious youth, aged 6-13, were randomly assigned to a family intervention program for childhood anxiety problems, which includes extensive parent communication training, or a child intervention program without parent-training. By comparing these two interventions, we tested if it was possible to improve parenting behaviors-such as intrusiveness-through intensive parent-training, above and beyond the effects of involving children in a child intervention program. We then tested the impact of this change in parental behaviors on children's ability to regulate fear and anxiety. We hypothesized that parent-training would reduce intrusiveness, which would in turn improve children's anxiety outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The child met DSM-IV criteria for a diagnosis of a principal anxiety disorder based on a semi-structured interview
* The child was not taking any psychiatric medication at the initial assessment, or was taking a stable dose of psychiatric medication (i.e., at least one month at a stable dose prior to the baseline assessment), and
* If medication was being used, families stated an intention to maintain that dose throughout the study.

Exclusion Criteria:

* The child was currently in child-focused psychotherapy
* The family was currently in family therapy or a parenting class
* Either the child or the parents evidenced psychotic symptoms
* The child began taking psychiatric medication or increased his/her dose of medication during the intervention, or
* For any reason the child or parents appeared unable to participate in the intervention program.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2000-03; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule--Child and Parent Versions | Posttreatment

SECONDARY OUTCOMES:
Multidimension Anxiety Scale for Children | Posttreatment

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Wood, Ph.D., Principal Investigator — University of California, Los Angeles; Marian Sigman, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Wood JJ, Piacentini JC, Southam-Gerow M, Chu BC, Sigman M. Family cognitive behavioral therapy for child anxiety disorders. J Am Acad Child Adolesc Psychiatry. 2006 Mar;45(3):314-321. doi: 10.1097/01.chi.0000196425.88341.b0. PMID 16540816